CLINICAL TRIAL: NCT03617965
Title: Mortality Due to Septic Shock Associated With Thrombocytopenia in the Intensive Care Unit
Brief Title: Mortality Due to Septic Shock Associated With Thrombocytopenia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidad de Guanajuato (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jaime Daniel Mondragón Uribe, Principal Investigator, Universidad de Guanajuato
Other Study IDs: UCISEP0718
Record Dates: First submitted 2018-07-23; First posted 2018-08-07 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Thrombocytopenia; Septic Shock; Sepsis Bacterial
MeSH Terms: conditions — Thrombocytopenia; Shock, Septic | interventions — Platelet Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mild thrombocytopenia: Patients with a platelet count of 100 × 10e9 to 149 × 10e9/L.
  Interventions: Diagnostic Test: Platelet count
- Moderate thrombocytopenia: Patients with a platelet count of 50 × 10e9 to 99 × 10e9/L
  Interventions: Diagnostic Test: Platelet count
- Severe thrombocytopenia: Patients with a platelet count<50 × 10e9/L
  Interventions: Diagnostic Test: Platelet count
- Control group: Patients with normal platelet count (i.e.150 × 10e9 to 399 × 10e9/L)
  Interventions: Diagnostic Test: Platelet count

INTERVENTIONS:
Diagnostic Test: Platelet count — All patients who are admitted to the intensive care unit of this hospital and meet the inclusion criteria will be followed for 90 days. There will be a complete review of the file that includes the entire hospitalization, in order to collect demographic information, clinical, laboratory reports, and imaging reports among others. Patients who are transferred to other units due to clinical improvement will be followed peripherally by the internal medicine department and the patients who are released due to clinical improvement will be contacted via telephone or in their next outpatient consultation with an internist.
  Other Names: Procalcitonin levels

SUMMARY:
A prospective longitudinal study similar to the one performed by Claushuis and colleagues (2016) will be performed in order to further understand the epidemiology and clinical relationship between platelet levels and mortality secondary to septic shock in a different population. The primary objective is to compare the mortality due to septic shock between patients with thrombocytopenia and patients with normal platelet levels in the ICU of the General Hospital of León, Gto. The secondary objectives are to identify the association between mortality due to septic shock and mild, moderate and severe thrombocytopenia in patients admitted to the ICU at 30, 60 and 90 days.

Research questions

Is there an association between thrombocytopenia and mortality due to septic shock in patients admitted to the critical medicine service? Our hypotheses are that:

1. Mortality from septic shock and thrombocytopenia at 30, 60 and 90 days will be higher in patients with thrombocytopenia than in patients normal platelet counts.

Is there an association between the degree of thrombocytopenia and mortality from septic shock in patients admitted to the critical medicine service? Our hypotheses are that:

1. Mortality from septic shock and thrombocytopenia at 30, 60 and 90 days will be higher in patients with mild thrombocytopenia than in patients without thrombocytopenia.
2. Mortality from septic shock and thrombocytopenia at 30, 60 and 90 days will be higher in patients with moderate thrombocytopenia than in patients without thrombocytopenia.
3. Mortality from septic shock and thrombocytopenia at 30, 60 and 90 days will be higher in patients with severe thrombocytopenia than in patients without thrombocytopenia.

DETAILED DESCRIPTION:
Background

Sepsis has a high morbidity and mortality, hence is a challenging medical problem throughout the world. Three therapeutic principles must be taken into account to improve organ dysfunction and survival in sepsis: 1) early and adequate antimicrobial therapy; 2) reestablishment of adequate tissue perfusion; and 3) timely identification and control of the septic foci. Moreover, survival in sepsis depends on the timely identification and appropriate treatment. Progressive advances in sepsis management over the past decades have led to reduced mortality indices. Mortality rates have decline progressively from 43% in 1993 to 37% in 2003, to 29% in 2007; furthermore, reaching a low in 2012 of 18.4%. All in all, in order to establish a global outlook and adequate therapeutic algorithms for sepsis, the factors associated with high mortality rates in septic shock must be identified.

Severe sepsis and septic shock are two clinical entities that have a great impact on intra-hospital morbidity and mortality, as well as on the cost of health care systems; accounting for a large proportion among the causes of admission to the intensive care unit (ICU). In the United States in 2013, septicemia was the hospital condition that accounted for the highest cost, reaching a total cost of $23.7 billion dollars (i.e. 6.2% of total hospitalization costs); followed by osteoarthritis (i.e. $16.5 billion dollars, 4.3% of total hospitalization costs), births (i.e. $13.3 billion, 3.5%), complications arising from medical devices, implants or grafts (i.e. $12.4 billion, 3.3%), and acute myocardial infarction (i.e. $12.1 billion, 3.2%).

The prevalence of sepsis at the ICU across multiple centers in Spain ranges between 6 and 30%. Furthermore, more than 50% of patients with sepsis develop severe sepsis and 25% septic shock. Carrillo-Esper and colleagues (2009) report that in Mexican public and private institutions, 27.3% of 40,957 hospitalizations (i.e. 11,183 cases) developed sepsis. This study which included data from ICUs of 24 out of 32 federal entities reports a mortality secondary to sepsis of 30.4%. In Mexico, the hospitalization costs of patients with sepsis is also a cause of concern, with a total estimated cost of $835 million dollars and an average patient cost of $73,000 dollars.

Sepsis definition

The systemic inflammatory response syndrome or SIRS response is the complex pathophysiological reaction to an insult (e.g. infection, trauma, burns). The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3), defines sepsis as a life-threatening organ dysfunction caused by a dysregulated host response to an infection. Severe sepsis is the sepsis complicated by organ dysfunction, which could progress to septic shock (i.e. sepsis-induced hypotension persisting despite adequate fluid resuscitation). The definitions for sepsis, septic shock, and organ dysfunction have essentially not changed in the past two decades. Despite its global importance, the recognition of sepsis is inadequate. Furthermore, the various manifestations of sepsis make diagnosis difficult, even for experienced physicians. Therefore, a comprehensive definition and clinical guidelines for sepsis management are needed; this would facilitate the clinical identification of sepsis by health professionals, thus improving the diagnostic accuracy and quantification of sepsis.

Thrombocytopenia

Platelets are the smallest blood cells, being only fragments of the megakaryocyte cytoplasm; however, they have a critical role in normal hemostasis and contribute to thrombotic disorders. The normal range of platelets in humans is 150,000-400,000 platelets per microliter of blood. The production of platelets is critically dependent on thrombopoietin, which acts on the differentiation and proliferation of megakaryocyte progenitors and in the maturation of megakaryocytes. Platelets have a short life of up to 10 days. Thrombocytopenia can be classified as: 1) mild, from 100 x 10^9 a 149 x 10^9/L; 2) moderate, from 50 x 10^9 to 99 x 10^9/L; and 3) severe, <50 x 10^9/L. It has been reported that 20% to 50% of patients in the ICU have thrombocytopenia. Aside from hemostatic functions and playing a central role in thrombosis, platelets participate in the immune response. Platelets react to an infectious agent by altering tissue integrity; contributing to the inflammatory cascade, as well as in the elimination process of pathogens and tissue repair. Platelets are activated in patients with SIRS and sepsis. Activation is followed by platelet isolation within the microcirculation and consequently giving rise to a thrombocytopenia. Platelets regulate inflammation and sepsis through multiple mechanisms. Among these mechanisms is innate immunity, where platelets express a receptor for lipopolysaccharide (LPS) Toll-like receptor-4, which contributes to thrombocytopenia through recruitment of neutrophils to the pulmonary system in a systemic response to LPS. Platelets also interact with other leukocytes, including monocytes. The interaction of activated platelets with monocytes induces the nuclear translocation of nuclear factor-kB (NF-kB) and expression of NF-kB dependent inflammatory genes. In addition to direct interactions with leukocytes, platelets contribute to inflammation and immune activation by releasing cytokines and cellular mediators stored in dense and alpha granules. The gold standard for the evaluation of thrombopoiesis is through bone marrow aspiration; however, since bone marrow aspiration is an invasive procedure, it is not frequently performed in clinical conditions such as sepsis.

The association between level of thrombocytopenia (i.e. mild, moderate, and severe) and mortality has been previously studied in sepsis. Claushuis and colleagues (2016), reported the mortality rates of 1,483 consecutive patients admitted to the intensive care unit with sepsis and degrees of thrombocytopenia (i.e. mild, moderate and severe, depending on platelet counts, very low <50 × 10^9/L, intermediate-low 50 × 10^9 to 99 × 10^9/L, low 100 × 10^9 to 149 × 10^9/L) against patients with normal platelet count (i.e. 150 × 10^9 to 399 × 10^9/L). The mortality reported at 30 days was 25.1%, 37.2%, and 54.1% for patients with mild, moderate and severe thrombocytopenia respectively. More studies are needed to confirm the relationship between the platelet levels and septic shock. We decided to conduct a prospective longitudinal study similar to the one performed by Claushuis and colleagues (2016) in our hospital in order to further understand the epidemiology and clinical relationship between platelet levels and mortality secondary to septic shock in a different population.

Complications: septic shock and multiple organ dysfunction

Sepsis can progress to septic shock, multiple organ failure and death if not recognized early. More than 50% of patients with sepsis develop severe sepsis and 25% septic shock; these figures represent 15% of all admissions to the ICU. Septic shock is defined as a septic process associated with circulatory, cellular and metabolic abnormalities; therefore, there is a higher risk of mortality compared to the unique presence of sepsis. Clinically, it includes patients who meet sepsis criteria and who, despite adequate fluid resuscitation, require vasopressors to maintain a mean arterial blood pressure (MAP) above 65mmHg and serum lactate concentration levels above 2 mmol/L. The factors that contribute to septic shock are 1) vasodilation; 2) endothelial dysfunction (i.e. increased permeability due to loss of vascular smooth muscle reactivity secondary to cellular and humoral mediators); 3) hypovolemia; and 4) bilateral ventricular dysfunction.

Multiple organ dysfunction (MOD) refers to progressive organic dysfunction in a severely ill patient; where homeostasis cannot be maintained without intervention. Because of its severity, the organic dysfunction is at one end of the spectrum of severity of the disease. Both infectious conditions (e.g. sepsis, septic shock), and non-infectious conditions (e.g. SIRS for pancreatitis) can present in MOD. MOD can manifest with affection to different systems such as: cardiovascular; pulmonary; hepatic; renal; gastrointestinal; and hematologic, among others. Multiple organ dysfunction can be defined as an increase of two or more points in the Sequential (Sepsis-Related) Organ Function Assessment score (SOFA). It is important to note that the SOFA score is a mark of organic dysfunction; consequently, it does not determine the individual treatment strategies, nor does it predict mortality according to demographic data (e.g. age) or the underlying conditions (e.g. stem cell transplant recipient, postoperative patient). However, the SOFA score helps identify those patients who potentially have a high risk of dying from an infection.

Singer and colleagues (2016) proposed the quickSOFA (qSOFA) scale in order to facilitate the identification of patients at risk of dying from sepsis. The qSOFA scale is a modified version of the SOFA scale, where a score greater than two points is associated with sepsis; consequently, having a poor prognosis. The qSOFA score can be easily calculated as it only has three components. Each component is assigned a point: 1) respiratory rate ≥22 ventilations per minute; 2) alteration of the mental state; and 3) systolic blood pressure ≤100mmHg). Hypoperfusion duration is directly associated with MOD, accounting for a mortality of 70%. According to SOFA score predictions, patients who meet these criteria for septic shock have a higher mortality than patients who do not meet the criteria (i.e. ≥40% versus ≥10%). Raith and colleagues (2017) report that in 182 ICUs in Australia and New Zeland, between 2000 and 2015, 184,875 patients were admitted with a primary admission diagnosis associated with an infectious process. The objective of the aforementioned study was to validate and evaluate the discriminatory capabilities of a two or more points increase in the SOFA score, a two or more increase in SIRS criteria, or a two or more points increase in the qSOFA score among critically ill patients with an infection. The retrospective study reported a greater capacity to predict the intra-hospital mortality of the SOFA scale over the SIRS criteria and qSOFA criteria.

Number of required patients and power calculation

The different sample sizes were calculated to detect statistically significant differences taking as parameters an α = 0.05 and with a statistical power of 0.8 (i.e. 1-β). The work carried out by Claushuis and colleagues (2016) was used to determine the minimum sample size needed to detect statistically significant changes using the categorical variables of mild, moderate and severe thrombocytopenia as previously defined in this protocol at 30, 60 and 90 days of stay in the ICU. The sample size calculator based on proportions of two samples considering the equality of the two extremes (i.e. tails of a Gaussian distribution), was used, available on the web page http://powerandsamplesize.com/. Table 8 summarizes the parameters used to perform these calculations. The parameters are the following: nA, number of patients with normal platelet concentration (i.e. higher than 150,000/μL and lower than 399,000/μL); nB, number of patients with thrombocytopenia; pA, mortality, in percentage, of patients with normal platelet concentration; pB, mortality, in percentage, of patients with thrombocytopenia; k (nA/nB), sampling proportion; N, sample size needed. Taking into account the results, we consider that a sample of more than 30 patients with severe thrombocytopenia is sufficient, while a sample of 105 patients with moderate thrombocytopenia is sufficient. A similar number of patients without thrombocytopenia is needed to make the comparative analysis of mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with sepsis (white blood cells >14,000μL) and thrombocytopenia (<150,000/μL).
* Patients who receive care in the ICU of the General Hospital of León, Gto.
* Patients with a complete file with 90-day evolution notes.

Exclusion Criteria:

* Patients diagnosed with cardiogenic, hypovolemic, anaphylactic and neurogenic shock
* Patients older than 80 years or younger than 18 years of age
* Patients referred from another ICU
* Patients with a diagnosis of neoplasia (i.e. hematologic and/or solid tumor)
* Pregnant women
* Patients with liver cirrhosis
* Patients with splenectomy
* Patients with thrombocytosis (i.e.> 400,000/μL) upon admission to ICU
* Patients with previous use of drugs that could produce thrombocytopenia ( e.g. calcium carbonate, acetylsalicylic acid, clopidogrel, dipyridamole, tamoxifen, cisplatin, bexarotene, doxorubicin, and lovastatin.

Elimination Criteria:

* Patients who do not have a follow-up at 30, 60 and 90 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the intensive care unit at the General Hospital of León, Guanajuato, Mexico. The sampling technique will be a convenience sampling as this is a regional urban hospital that serves a total population of approximately 1.5 million people.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival and mortality rate | 30 days after ICU admission
  Multivariate-adjusted Cox proportional hazards regression models will be used to study the relationship between the diagnostic groups upon admission to the ICU and the mortality rate. Cox regression models adjusted to control the influence of sociodemographic variables will be used. Kaplan-Meier graphs will be used to show differences in the risk of progression to sepsis, septic shock, and death at 30 days.

SECONDARY OUTCOMES:
Survival and mortality rate | 60 days after ICU admission
  Multivariate-adjusted Cox proportional hazards regression models will be used to study the relationship between the diagnostic groups upon admission to the ICU and the mortality rate. Cox regression models adjusted to control the influence of sociodemographic variables will be used. Kaplan-Meier graphs will be used to show differences in the risk of progression to sepsis, septic shock, and death at 60 days.
Survival and mortality rate | 90 days after ICU admission
  Multivariate-adjusted Cox proportional hazards regression models will be used to study the relationship between the diagnostic groups upon admission to the ICU and the mortality rate. Cox regression models adjusted to control the influence of sociodemographic variables will be used. Kaplan-Meier graphs will be used to show differences in the risk of progression to sepsis, septic shock, and death at 90 days.
Association between platelet levels and diagnosis | 30 days after ICU admission
  Will be evaluated using a principal component analysis.
Platelet serum levels will be compared with the different clinical outcomes | 30 days after ICU admission
  The potentially associated variables will be added through the analysis of covariance (ANCOVA) or linear regression adjusted for age, sex, and diagnosis depending on the most appropriate model to assess the prognostic factors to develop sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime D Mondragón, MD, MS, Principal Investigator — University Medical Center Groningen
Locations (1):
- Hospital General de León, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No
Abiding by the Declaration of Helsinki, patient anonymity will be guaranteed.

REFERENCES:
- [Result] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Result] Armstrong BA, Betzold RD, May AK. Sepsis and Septic Shock Strategies. Surg Clin North Am. 2017 Dec;97(6):1339-1379. doi: 10.1016/j.suc.2017.07.003. Epub 2017 Oct 5. PMID 29132513
- [Result] Asaduzzaman M, Lavasani S, Rahman M, Zhang S, Braun OO, Jeppsson B, Thorlacius H. Platelets support pulmonary recruitment of neutrophils in abdominal sepsis. Crit Care Med. 2009 Apr;37(4):1389-96. doi: 10.1097/CCM.0b013e31819ceb71. PMID 19242347
- [Result] Balk RA. Systemic inflammatory response syndrome (SIRS): where did it come from and is it still relevant today? Virulence. 2014 Jan 1;5(1):20-6. doi: 10.4161/viru.27135. Epub 2013 Nov 13. PMID 24280933
- [Result] Bassetti M, Righi E, Ansaldi F, Merelli M, Trucchi C, De Pascale G, Diaz-Martin A, Luzzati R, Rosin C, Lagunes L, Trecarichi EM, Sanguinetti M, Posteraro B, Garnacho-Montero J, Sartor A, Rello J, Rocca GD, Antonelli M, Tumbarello M. A multicenter study of septic shock due to candidemia: outcomes and predictors of mortality. Intensive Care Med. 2014 Jun;40(6):839-45. doi: 10.1007/s00134-014-3310-z. Epub 2014 May 8. PMID 24807083
- [Result] Blair P, Flaumenhaft R. Platelet alpha-granules: basic biology and clinical correlates. Blood Rev. 2009 Jul;23(4):177-89. doi: 10.1016/j.blre.2009.04.001. Epub 2009 May 17. PMID 19450911
- [Result] Boehme AK, Ranawat P, Luna J, Kamel H, Elkind MS. Risk of Acute Stroke After Hospitalization for Sepsis: A Case-Crossover Study. Stroke. 2017 Mar;48(3):574-580. doi: 10.1161/STROKEAHA.116.016162. Epub 2017 Feb 14. PMID 28196938
- [Result] Brun-Buisson C. The epidemiology of the systemic inflammatory response. Intensive Care Med. 2000;26 Suppl 1(Suppl 1):S64-74. doi: 10.1007/s001340051121. PMID 10786961
- [Result] Carrillo-Esper R, Carrillo-Cordova JR, Carrillo-Cordova LD. Epidemiological study of sepsis in Mexican intensive care units. Cir Cir. 2009 Jul-Aug;77(4):301-8; 279-85. English, Spanish. PMID 19919792
- [Result] Casserly B, Phillips GS, Schorr C, Dellinger RP, Townsend SR, Osborn TM, Reinhart K, Selvakumar N, Levy MM. Lactate measurements in sepsis-induced tissue hypoperfusion: results from the Surviving Sepsis Campaign database. Crit Care Med. 2015 Mar;43(3):567-73. doi: 10.1097/CCM.0000000000000742. PMID 25479113
- [Result] Churpek MM, Snyder A, Han X, Sokol S, Pettit N, Howell MD, Edelson DP. Quick Sepsis-related Organ Failure Assessment, Systemic Inflammatory Response Syndrome, and Early Warning Scores for Detecting Clinical Deterioration in Infected Patients outside the Intensive Care Unit. Am J Respir Crit Care Med. 2017 Apr 1;195(7):906-911. doi: 10.1164/rccm.201604-0854OC. PMID 27649072
- [Result] Clark SR, Ma AC, Tavener SA, McDonald B, Goodarzi Z, Kelly MM, Patel KD, Chakrabarti S, McAvoy E, Sinclair GD, Keys EM, Allen-Vercoe E, Devinney R, Doig CJ, Green FH, Kubes P. Platelet TLR4 activates neutrophil extracellular traps to ensnare bacteria in septic blood. Nat Med. 2007 Apr;13(4):463-9. doi: 10.1038/nm1565. Epub 2007 Mar 25. PMID 17384648
- [Result] Claushuis TA, van Vught LA, Scicluna BP, Wiewel MA, Klein Klouwenberg PM, Hoogendijk AJ, Ong DS, Cremer OL, Horn J, Franitza M, Toliat MR, Nurnberg P, Zwinderman AH, Bonten MJ, Schultz MJ, van der Poll T; Molecular Diagnosis and Risk Stratification of Sepsis Consortium. Thrombocytopenia is associated with a dysregulated host response in critically ill sepsis patients. Blood. 2016 Jun 16;127(24):3062-72. doi: 10.1182/blood-2015-11-680744. Epub 2016 Mar 8. PMID 26956172
- [Result] Clec'h C, Fosse JP, Karoubi P, Vincent F, Chouahi I, Hamza L, Cupa M, Cohen Y. Differential diagnostic value of procalcitonin in surgical and medical patients with septic shock. Crit Care Med. 2006 Jan;34(1):102-7. doi: 10.1097/01.ccm.0000195012.54682.f3. PMID 16374163
- [Result] Cloutier N, Pare A, Farndale RW, Schumacher HR, Nigrovic PA, Lacroix S, Boilard E. Platelets can enhance vascular permeability. Blood. 2012 Aug 9;120(6):1334-43. doi: 10.1182/blood-2012-02-413047. Epub 2012 Apr 27. PMID 22544703
- [Result] Danai PA, Moss M, Mannino DM, Martin GS. The epidemiology of sepsis in patients with malignancy. Chest. 2006 Jun;129(6):1432-40. doi: 10.1378/chest.129.6.1432. PMID 16778259
- [Result] de Oliveira FS, Freitas FG, Ferreira EM, de Castro I, Bafi AT, de Azevedo LC, Machado FR. Positive fluid balance as a prognostic factor for mortality and acute kidney injury in severe sepsis and septic shock. J Crit Care. 2015 Feb;30(1):97-101. doi: 10.1016/j.jcrc.2014.09.002. Epub 2014 Sep 6. PMID 25269788
- [Result] De Silva E, Kim H. Drug-induced thrombocytopenia: Focus on platelet apoptosis. Chem Biol Interact. 2018 Mar 25;284:1-11. doi: 10.1016/j.cbi.2018.01.015. Epub 2018 Feb 2. PMID 29410286
- [Result] Deutsch VR, Tomer A. Advances in megakaryocytopoiesis and thrombopoiesis: from bench to bedside. Br J Haematol. 2013 Jun;161(6):778-93. doi: 10.1111/bjh.12328. Epub 2013 Apr 18. PMID 23594368
- [Result] Dewitte A, Lepreux S, Villeneuve J, Rigothier C, Combe C, Ouattara A, Ripoche J. Blood platelets and sepsis pathophysiology: A new therapeutic prospect in critically [corrected] ill patients? Ann Intensive Care. 2017 Dec 1;7(1):115. doi: 10.1186/s13613-017-0337-7. PMID 29192366
- [Result] Dremsizov T, Clermont G, Kellum JA, Kalassian KG, Fine MJ, Angus DC. Severe sepsis in community-acquired pneumonia: when does it happen, and do systemic inflammatory response syndrome criteria help predict course? Chest. 2006 Apr;129(4):968-78. doi: 10.1378/chest.129.4.968. PMID 16608946
- [Result] Esposito S, De Simone G, Boccia G, De Caro F, Pagliano P. Sepsis and septic shock: New definitions, new diagnostic and therapeutic approaches. J Glob Antimicrob Resist. 2017 Sep;10:204-212. doi: 10.1016/j.jgar.2017.06.013. Epub 2017 Jul 22. PMID 28743646
- [Result] Fujishima S. Organ dysfunction as a new standard for defining sepsis. Inflamm Regen. 2016 Nov 15;36:24. doi: 10.1186/s41232-016-0029-y. eCollection 2016. PMID 29259697
- [Result] George JN. Platelets. Lancet. 2000 Apr 29;355(9214):1531-9. doi: 10.1016/S0140-6736(00)02175-9. PMID 10801186
- [Result] Girard TD, Opal SM, Ely EW. Insights into severe sepsis in older patients: from epidemiology to evidence-based management. Clin Infect Dis. 2005 Mar 1;40(5):719-27. doi: 10.1086/427876. Epub 2005 Jan 28. PMID 15714419
- [Result] Greco E, Lupia E, Bosco O, Vizio B, Montrucchio G. Platelets and Multi-Organ Failure in Sepsis. Int J Mol Sci. 2017 Oct 20;18(10):2200. doi: 10.3390/ijms18102200. PMID 29053592
- [Result] Gupta S, Sakhuja A, Kumar G, McGrath E, Nanchal RS, Kashani KB. Culture-Negative Severe Sepsis: Nationwide Trends and Outcomes. Chest. 2016 Dec;150(6):1251-1259. doi: 10.1016/j.chest.2016.08.1460. Epub 2016 Sep 9. PMID 27615024
- [Result] Hara T, Shimizu K, Ogawa F, Yanaba K, Iwata Y, Muroi E, Takenaka M, Komura K, Hasegawa M, Fujimoto M, Sato S. Platelets control leukocyte recruitment in a murine model of cutaneous arthus reaction. Am J Pathol. 2010 Jan;176(1):259-69. doi: 10.2353/ajpath.2010.081117. Epub 2009 Dec 11. PMID 20008131
- [Result] Haas SA, Lange T, Saugel B, Petzoldt M, Fuhrmann V, Metschke M, Kluge S. Severe hyperlactatemia, lactate clearance and mortality in unselected critically ill patients. Intensive Care Med. 2016 Feb;42(2):202-10. doi: 10.1007/s00134-015-4127-0. Epub 2015 Nov 10. PMID 26556617
- [Result] Herran-Monge R, Muriel-Bombin A, Garcia-Garcia MM, Merino-Garcia PA, Martinez-Barrios M, Andaluz D, Ballesteros JC, Dominguez-Berrot AM, Moradillo-Gonzalez S, Macias S, Alvarez-Martinez B, Fernandez-Calavia MJ, Tarancon C, Villar J, Blanco J. Epidemiology and Changes in Mortality of Sepsis After the Implementation of Surviving Sepsis Campaign Guidelines. J Intensive Care Med. 2019 Sep;34(9):740-750. doi: 10.1177/0885066617711882. Epub 2017 Jun 26. PMID 28651474
- [Result] Hollenberg SM. Inotrope and vasopressor therapy of septic shock. Crit Care Nurs Clin North Am. 2011 Mar;23(1):127-48. doi: 10.1016/j.ccell.2010.12.008. PMID 21316572
- [Result] Jones GR, Lowes JA. The systemic inflammatory response syndrome as a predictor of bacteraemia and outcome from sepsis. QJM. 1996 Jul;89(7):515-22. doi: 10.1093/qjmed/89.7.515. PMID 8759492
- [Result] Klein Klouwenberg PM, Frencken JF, Kuipers S, Ong DS, Peelen LM, van Vught LA, Schultz MJ, van der Poll T, Bonten MJ, Cremer OL; MARS Consortium *. Incidence, Predictors, and Outcomes of New-Onset Atrial Fibrillation in Critically Ill Patients with Sepsis. A Cohort Study. Am J Respir Crit Care Med. 2017 Jan 15;195(2):205-211. doi: 10.1164/rccm.201603-0618OC. PMID 27467907
- [Result] Knaus WA, Sun X, Nystrom O, Wagner DP. Evaluation of definitions for sepsis. Chest. 1992 Jun;101(6):1656-62. doi: 10.1378/chest.101.6.1656. PMID 1600787
- [Result] Koyama K, Katayama S, Muronoi T, Tonai K, Goto Y, Koinuma T, Shima J, Nunomiya S. Time course of immature platelet count and its relation to thrombocytopenia and mortality in patients with sepsis. PLoS One. 2018 Jan 30;13(1):e0192064. doi: 10.1371/journal.pone.0192064. eCollection 2018. PMID 29381746
- [Result] Kreger BE, Craven DE, McCabe WR. Gram-negative bacteremia. IV. Re-evaluation of clinical features and treatment in 612 patients. Am J Med. 1980 Mar;68(3):344-55. doi: 10.1016/0002-9343(80)90102-3. PMID 6987871
- [Result] Martin GS, Mannino DM, Moss M. The effect of age on the development and outcome of adult sepsis. Crit Care Med. 2006 Jan;34(1):15-21. doi: 10.1097/01.ccm.0000194535.82812.ba. PMID 16374151
- [Result] Marshall JC, Cook DJ, Christou NV, Bernard GR, Sprung CL, Sibbald WJ. Multiple organ dysfunction score: a reliable descriptor of a complex clinical outcome. Crit Care Med. 1995 Oct;23(10):1638-52. doi: 10.1097/00003246-199510000-00007. PMID 7587228
- [Result] Minasyan H. Sepsis and septic shock: Pathogenesis and treatment perspectives. J Crit Care. 2017 Aug;40:229-242. doi: 10.1016/j.jcrc.2017.04.015. Epub 2017 Apr 18. PMID 28448952
- [Result] Netea MG, van der Meer JW. Immunodeficiency and genetic defects of pattern-recognition receptors. N Engl J Med. 2011 Jan 6;364(1):60-70. doi: 10.1056/NEJMra1001976. No abstract available. PMID 21208109
- [Result] Nduka OO, Parrillo JE. The pathophysiology of septic shock. Crit Care Nurs Clin North Am. 2011 Mar;23(1):41-66. doi: 10.1016/j.ccell.2010.12.003. PMID 21316567
- [Result] O'Brien JM Jr, Lu B, Ali NA, Martin GS, Aberegg SK, Marsh CB, Lemeshow S, Douglas IS. Alcohol dependence is independently associated with sepsis, septic shock, and hospital mortality among adult intensive care unit patients. Crit Care Med. 2007 Feb;35(2):345-50. doi: 10.1097/01.CCM.0000254340.91644.B2. PMID 17205003
- [Result] Peres Bota D, Lopes Ferreira F, Melot C, Vincent JL. Body temperature alterations in the critically ill. Intensive Care Med. 2004 May;30(5):811-6. doi: 10.1007/s00134-004-2166-z. Epub 2004 Feb 4. PMID 15127194
- [Result] Poutsiaka DD, Davidson LE, Kahn KL, Bates DW, Snydman DR, Hibberd PL. Risk factors for death after sepsis in patients immunosuppressed before the onset of sepsis. Scand J Infect Dis. 2009;41(6-7):469-79. doi: 10.1080/00365540902962756. PMID 19452348
- [Result] Prescott HC, Dickson RP, Rogers MA, Langa KM, Iwashyna TJ. Hospitalization Type and Subsequent Severe Sepsis. Am J Respir Crit Care Med. 2015 Sep 1;192(5):581-8. doi: 10.1164/rccm.201503-0483OC. PMID 26016947
- [Result] Raith EP, Udy AA, Bailey M, McGloughlin S, MacIsaac C, Bellomo R, Pilcher DV; Australian and New Zealand Intensive Care Society (ANZICS) Centre for Outcomes and Resource Evaluation (CORE). Prognostic Accuracy of the SOFA Score, SIRS Criteria, and qSOFA Score for In-Hospital Mortality Among Adults With Suspected Infection Admitted to the Intensive Care Unit. JAMA. 2017 Jan 17;317(3):290-300. doi: 10.1001/jama.2016.20328. PMID 28114553
- [Result] Ruiz-Alvarez MJ, Garcia-Valdecasas S, De Pablo R, Sanchez Garcia M, Coca C, Groeneveld TW, Roos A, Daha MR, Arribas I. Diagnostic efficacy and prognostic value of serum procalcitonin concentration in patients with suspected sepsis. J Intensive Care Med. 2009 Jan-Feb;24(1):63-71. doi: 10.1177/0885066608327095. Epub 2008 Dec 2. PMID 19054806
- [Result] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Result] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Result] Russell JA, Rush B, Boyd J. Pathophysiology of Septic Shock. Crit Care Clin. 2018 Jan;34(1):43-61. doi: 10.1016/j.ccc.2017.08.005. PMID 29149941
- [Result] Schuetz P, Birkhahn R, Sherwin R, Jones AE, Singer A, Kline JA, Runyon MS, Self WH, Courtney DM, Nowak RM, Gaieski DF, Ebmeyer S, Johannes S, Wiemer JC, Schwabe A, Shapiro NI. Serial Procalcitonin Predicts Mortality in Severe Sepsis Patients: Results From the Multicenter Procalcitonin MOnitoring SEpsis (MOSES) Study. Crit Care Med. 2017 May;45(5):781-789. doi: 10.1097/CCM.0000000000002321. PMID 28257335
- [Result] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- [Result] Shorr AF, Tabak YP, Killian AD, Gupta V, Liu LZ, Kollef MH. Healthcare-associated bloodstream infection: A distinct entity? Insights from a large U.S. database. Crit Care Med. 2006 Oct;34(10):2588-95. doi: 10.1097/01.CCM.0000239121.09533.09. PMID 16915117
- [Result] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Tang Y, Choi J, Kim D, Tudtud-Hans L, Li J, Michel A, Baek H, Hurlow A, Wang C, Nguyen HB. Clinical predictors of adverse outcome in severe sepsis patients with lactate 2-4 mM admitted to the hospital. QJM. 2015 Apr;108(4):279-87. doi: 10.1093/qjmed/hcu186. Epub 2014 Sep 4. PMID 25193540
- [Result] Tang BM, Eslick GD, Craig JC, McLean AS. Accuracy of procalcitonin for sepsis diagnosis in critically ill patients: systematic review and meta-analysis. Lancet Infect Dis. 2007 Mar;7(3):210-7. doi: 10.1016/S1473-3099(07)70052-X. PMID 17317602
- [Result] Theerawit P, Na Petvicharn C, Tangsujaritvijit V, Sutherasan Y. The Correlation Between Arterial Lactate and Venous Lactate in Patients With Sepsis and Septic Shock. J Intensive Care Med. 2018 Feb;33(2):116-120. doi: 10.1177/0885066616663169. Epub 2016 Aug 8. PMID 27502951
- [Result] Thiery-Antier N, Binquet C, Vinault S, Meziani F, Boisrame-Helms J, Quenot JP; EPIdemiology of Septic Shock Group. Is Thrombocytopenia an Early Prognostic Marker in Septic Shock? Crit Care Med. 2016 Apr;44(4):764-72. doi: 10.1097/CCM.0000000000001520. PMID 26670473
- [Result] Tolsma V, Schwebel C, Azoulay E, Darmon M, Souweine B, Vesin A, Goldgran-Toledano D, Lugosi M, Jamali S, Cheval C, Adrie C, Kallel H, Descorps-Declere A, Garrouste-Orgeas M, Bouadma L, Timsit JF. Sepsis severe or septic shock: outcome according to immune status and immunodeficiency profile. Chest. 2014 Nov;146(5):1205-1213. doi: 10.1378/chest.13-2618. PMID 25033349
- [Result] Torio CM, Moore BJ. National Inpatient Hospital Costs: The Most Expensive Conditions by Payer, 2013. 2016 May. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #204. Available from http://www.ncbi.nlm.nih.gov/books/NBK368492/ PMID 27359025
- [Result] van Vught LA, Wiewel MA, Klein Klouwenberg PM, Hoogendijk AJ, Scicluna BP, Ong DS, Cremer OL, Horn J, Bonten MM, Schultz MJ, van der Poll T; Molecular Diagnosis and Risk Stratification of Sepsis Consortium. Admission Hyperglycemia in Critically Ill Sepsis Patients: Association With Outcome and Host Response. Crit Care Med. 2016 Jul;44(7):1338-46. doi: 10.1097/CCM.0000000000001650. PMID 26958752
- [Result] Vincent JL, Bihari DJ, Suter PM, Bruining HA, White J, Nicolas-Chanoin MH, Wolff M, Spencer RC, Hemmer M. The prevalence of nosocomial infection in intensive care units in Europe. Results of the European Prevalence of Infection in Intensive Care (EPIC) Study. EPIC International Advisory Committee. JAMA. 1995 Aug 23-30;274(8):639-44. PMID 7637145
- [Result] Wang B, Chen G, Cao Y, Xue J, Li J, Wu Y. Correlation of lactate/albumin ratio level to organ failure and mortality in severe sepsis and septic shock. J Crit Care. 2015 Apr;30(2):271-5. doi: 10.1016/j.jcrc.2014.10.030. Epub 2014 Nov 11. PMID 25537574
- [Result] Walkey AJ, Wiener RS, Ghobrial JM, Curtis LH, Benjamin EJ. Incident stroke and mortality associated with new-onset atrial fibrillation in patients hospitalized with severe sepsis. JAMA. 2011 Nov 23;306(20):2248-54. doi: 10.1001/jama.2011.1615. Epub 2011 Nov 13. PMID 22081378
- [Result] Williamson DR, Albert M, Heels-Ansdell D, Arnold DM, Lauzier F, Zarychanski R, Crowther M, Warkentin TE, Dodek P, Cade J, Lesur O, Lim W, Fowler R, Lamontagne F, Langevin S, Freitag A, Muscedere J, Friedrich JO, Geerts W, Burry L, Alhashemi J, Cook D; PROTECT collaborators, the Canadian Critical Care Trials Group, and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Thrombocytopenia in critically ill patients receiving thromboprophylaxis: frequency, risk factors, and outcomes. Chest. 2013 Oct;144(4):1207-1215. doi: 10.1378/chest.13-0121. PMID 23788287
- [Result] Zahar JR, Timsit JF, Garrouste-Orgeas M, Francais A, Vesin A, Descorps-Declere A, Dubois Y, Souweine B, Haouache H, Goldgran-Toledano D, Allaouchiche B, Azoulay E, Adrie C. Outcomes in severe sepsis and patients with septic shock: pathogen species and infection sites are not associated with mortality. Crit Care Med. 2011 Aug;39(8):1886-95. doi: 10.1097/CCM.0b013e31821b827c. PMID 21516036